CLINICAL TRIAL: NCT04577144
Title: Remission From Chronic Opioid Use: Study of Environmental and Socioeconomic Factors on Recovery - Long Term
Brief Title: An Observational Study of Environmental and Socioeconomic Factors in Opioid Recovery - Long Term
Acronym: RECOVER-LT
Status: Terminated | Type: Observational
Why Stopped: Study re-scoped due to COVID-19 pandemic.
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: INDV-6000-H03
Record Dates: First submitted 2020-09-18; First posted 2020-10-06 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals who participated in the RECOVER study: Individuals who enrolled in the Remission from Chronic Opioid Use-Studying Environmental and Socio-Economic Factors on Recovery (RECOVER) study. Individuals who received at least one injection in a SUBLOCADE Phase III program were eligible to participate in the original study.
  Interventions: Other: Online survey only

INTERVENTIONS:
Other: Online survey only — There are no interventions planned for this study. This is an observational study only.

SUMMARY:
The purpose of this study (RECOVER-LT) is to better understand the long-term paths of recovery from opioid use disorder (OUD) for an additional 5 year period after the original RECOVER (NCT03604861) study. Long-term patterns of abstinence/opioid misuse as well as measures of participants' physical, psychological, social and economic well being will be monitored in order to identify factors associated with recovery from OUD.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who enrolled in the RECOVER study
* Ability to comply with current study protocol requirements for data collection
* Provide informed consent

Exclusion Criteria:

* Minors will not be included
* Prisoners will not be included. If participants become incarcerated during this study, they will not be contacted to complete assessments during their incarceration. If the incarceration ends during the study, they may be contacted to participate in assessments
* Adults who are not capable of consenting on their own behalf

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from individuals who enrolled in the RECOVER study
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Abstinence from opioid use | Change from baseline after a period of up to 5 years will be reported.
  Self-reported 7-day point prevalence of opioid use will be measured approximately every 4 months
Abstinence from opioid use | Change from baseline after a period of up to 5 years will be reported.
  Self-reported 30-day point prevalence of opioid use will be measured approximately every 4 months
Abstinence from opioid use | Change from baseline after a period of up to 5 years will be reported.
  Self-reported opioid use in the time period since last assessment will be measured approximately every 4 months

SECONDARY OUTCOMES:
Recovery from opioid use disorder (OUD) | Up to 14 assessments approximately every 4 months from Assessment 1 to Assessment 14 over a period of up to 5 years.
  Assessment of recovery will include assessment of symptoms of OUD as measured by Subjective Opiate Withdrawal Scale (SOWS). Higher numbers indicate worse outcomes
Recovery from opioid use disorder (OUD) | Up to 14 assessments approximately every 4 months from Assessment 1 to Assessment 14 over a period of up to 5 years
  Assessment of recovery will include assessment of symptoms of OUD as measured by an Opioid Craving Scale, using a visual analog scale which measures moment opioid craving, craving over the past 7 days and craving if participant was present in a previous drug use environment. Higher numbers indicate worse symptoms of craving.
Quality of life measures-household chaos: CHAOS | Up to 14 assessments approximately every 4 months from Assessment 1 to Assessment 14 over a period of up to 5 years
  Measured by CHAOS, the Confusion, hubbub and order scale-short form. This is a 6-item scale which uses yes-no questions to measure the amount of household disorder. Higher levels of household disorder are associated with worse outcomes.
Satisfaction with medications received to treat OUD: Medication Satisfaction Questionnaire | Measured annually from Assessment 1 to Assessment 14 over a period of up to 5 years
  Completion of a Medication Satisfaction Questionnaire for those receiving medication to treat OUD
Assessment of recovery and treatment | Measured annually from Assessment 1 to Assessment 14 over a period of up to 5 years
  Completion of a Treatment Effectiveness Assessment, a patient-centered instrument for evaluating progress in recovery from addiction. Patients provide both numerical responses and representative details on their substance use, health, lifestyle, and community.
Recovery from opioid use disorder (OUD) | Measured annually from Assessment 1 to Assessment 14 over a period of up to 5 years
  Participants will be asked to complete a self-assessment of recovery. Participants will rate their perceived success in recovery qualitatively
Assessment of functional impairment | Up to 14 assessments approximately every 4 months from Assessment 1 to Assessment 14 over a period of up to 5 years
  Measured by completion of the Sheehan Disability Scale, which is a 5-item self-report tool that assesses functional impairment in work/school, social life, and family life. Scores range from 0-30, and higher scores indicate worse impairment.
Quality of life-depression: Beck Depression Inventory-II | Up to 14 assessments approximately every 4 months from Assessment 1 to Assessment 14 over a period of up to 5 years
  Measured by the Beck Depression Inventory-II which measures characteristic attitudes and symptoms of depression. Scores can range from 0-63 and higher numbers indicate worse symptoms of depression.
Quality of life measures - broad domains: WHOQOL-BREF | Up to 14 assessments approximately every 4 months from Assessment 1 to Assessment 14 over a period of up to 5 years
  Measured by the World Health Organization Quality of Life Assessment - Abbreviated Version(WHOQOL-BREF) which measures physical health, social relationships, psychological health and environment
Quality of life measures-overall: Medical Outcomes Study, Short-Form- 12 (SF-12) | Up to 14 assessments approximately every 4 months from Assessment 1 to Assessment 14 over a period of up to 5 years
  Measured by the 12 Item Short Form Health Survey (SF-12) which assesses mental and physical functioning and overall health-related quality of life over a period of time.
Quality of life measures-pain: Brief Pain Inventory | Up to 14 assessments approximately every 4 months from Assessment 1 to Assessment 14 over a period of up to 5 years
  Measured by the Brief Pain Inventory which rates pain severity
Quality of life measures-adverse experiences: Holmes-Rahe Life Stress Inventory | Up to 14 assessments approximately every 4 months from Assessment 1 to Assessment 14 over a period of up to 5 years
  Measured by the Holmes-Rahe Life Stress Inventory which lists stressful life events that could contribute to illness. Higher scores indicate an increased susceptibility to stress-related health breakdown
Number of crimes committed | Up to 14 assessments approximately every 4 months from Assessment 1 to Assessment 14 over a period of up to 5 years
  Participants will complete surveys to identify the number and type of criminal incidents in the time period since last assessment
Occurrence of overdose | Up to 14 assessments from Assessment 1 to Assessment 14 over a period of up to 5 years
  Participants will complete survey to identify if an overdose occurred and the number of times of an overdose in the time period since last assessment
Hospitalization and urgent care utilization | Up to 14 assessments from Assessment 1 to Assessment 14 over a period of up to 5 years
  Participants will complete survey to identify if hospitals and emergency room visits occurred and the frequency of visits to the hospitals and emergency rooms in the time period since last assessment

CONTACTS AND LOCATIONS:
Overall Officials: Warren Bickel, Principal Investigator — Virginia Tech Carilion
Locations (1):
- Addiction Recovery Research Center and Fralin Biomedical Research Institute, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Craft WH, Tegge AN, Keith DR, Shin H, Williams J, Athamneh LN, Stein JS, Chilcoat HD, Le Moigne A, DeVeaugh-Geiss A, Bickel WK. Recovery from opioid use disorder: A 4-year post-clinical trial outcomes study. Drug Alcohol Depend. 2022 May 1;234:109389. doi: 10.1016/j.drugalcdep.2022.109389. Epub 2022 Mar 9. PMID 35287034
- [Derived] Keith DR, Tegge AN, Stein JS, Athamneh LN, Craft WH, Chilcoat HD, Le Moigne A, DeVeaugh-Geiss A, Bickel WK. Struggling With Recovery From Opioids: Who Is at Risk During COVID-19? J Addict Med. 2023 May-Jun 01;17(3):e156-e163. doi: 10.1097/ADM.0000000000001096. Epub 2022 Oct 16. PMID 37267169
- See also: Recovery from opioid use disorder: A 4-year post-clinical trial outcomes study — https://pubmed.ncbi.nlm.nih.gov/35287034/